CLINICAL TRIAL: NCT00568542
Title: Pilot Study to Assess the Effect of Low Dose Epoetin Beta Administered for Six Month in Patients With Ischemic Heart Failure Subjected to Percutaneous Coronary Intervention (PCI)
Brief Title: Chronic, Low Dose Erythropoetin Beta in Ischemic Cardiomyopathy
Acronym: EPOHeart
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Priv.-Doz. Dr. Martin W. Bergmann, Charité Campus Buch, University Medicine Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 8514077463; EudraCT number 2004-002646-35; EK 6 EA 3/015/05; KP-3910-4030711
Record Dates: First submitted 2007-12-05; First posted 2007-12-06 (Estimated); Last update posted 2009-08-04 (Estimated); Status verified 2009-08

CONDITIONS: Ischemic Cardiomyopathy
Keywords: cardiomyopathy; ischemia; percutaneous coronary intervention; remodeling
MeSH Terms: conditions — Cardiomyopathies; Ischemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): 35 I.E. erythropoetin beta given by subcutaneous injection once per week for 6 months. The drug is self-administered.
  Interventions: Drug: erythropoetin beta
- 2 (Placebo Comparator): Placebo to erythropoetin beta.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: erythropoetin beta — 35 I.E. kg body weight subcutaneous once per week for 6 months
  Other Names: NeoRecormom 10.000 I.E. Patronen Zul.Nr. EU/1/97/031/021-022
  Arms: 1
Drug: placebo — 35 I.E. kg body weight placebo to erythropoetin beta
  Other Names: Placebo to NeoRecormon 10.000 patron
  Arms: 2

SUMMARY:
The study is testing the hypothesis, that the application of low dose erythropoetin beta (35 I.E./kg BW/week) for 6 months following successful coronary revascularization by PCI improves left ventricular remodeling as assessed by cardiac MRI.

DETAILED DESCRIPTION:
Several effects known to be exerted by erythropoetin (EPO) directly in the heart independent of hemoglobin levels could be of value immediately after revascularization procedures in ischemic cardiac remodeling: the generation of new capillaries is enhanced by the mobilization of endothelial progenitor cells from the bone marrow. EPO is neuron- and cardio-protective after ischemia/reperfusion. Administration of EPO enhances neuronal progenitors to differentiate into functional neurons; this observation may also be valid for the cardiac compartment. The concept of organ-specific effects of EPO independent of hemoglobin levels is supported by the analysis of EPO analogues lacking hematopoietic activity. In humans, currently this concept can only be tested by the use of EPO-doses that do not affect hemoglobin levels. The concept is valid as clinical trials have been performed showing that doses as low as 5000 I.U. EPO once weekly increase the levels of endothelial progenitor cells in blood. On the other hand, recent clinical trials have also shown neutral or even deleterious effects of high dose EPO treatment raising hemoglobin levels to above 12mg/dl in pre-dialysis patients concerning cardiovascular endpoints. Therefore, the chronic, hemoglobin-neutral administration of low doses of EPO might be a successful approach concerning ischemic cardiomyopathy.

Study outline:

This investigator initiated, double-blind, placebo-controlled study is testing the hypothesis, that low doses of erythropoietin beta (35 I.U./kg body weight) started within 14 days after a successful percutaneous coronary intervention enhance left ventricular remodeling as determined by comparison of two cardiac MRI´s over a course of 6 months. Secondary endpoints include changes in diastolic dysfunction as measured by echocardiography, VO2 measured by spiroergometry and serum brain natriuretic peptide levels.

ELIGIBILITY:
Inclusion Criteria:

* successful coronary intervention < 14 days
* regional contraction deficit of the left ventricle as detected either by echocardiography or cardiacMRI
* globally reduced ejection fraction (cardiac MRI or echocardiography: < 60%)
* willing and able to cooperate
* voluntary participation

Exclusion Criteria:

* contraindication for cardiac MRI (i.e. pacemaker, ICD current or within the next 6 months, other metal implants)
* cardiogenic shock at time of inclusion
* uncontrolled hypertension (systolic blood pressure > 180mmHg)
* hemoglobin > 16mg/dl
* thrombocytosis
* malignant tumor
* missing informed consent
* renal failure (creatinine > 300 mg/dl)
* liver failure
* other prognosis limiting, severe diseases (i.e. dementia)
* indication for open label erythropoietin treatment
* allergy towards solvents of the EPO preparation
* woman of childbearing potential
* other clinical study within the preceding 30days
* known alcohol or drug abuse
* neurologic or psychiatry disorders
* previous organ transplantation

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2006-05; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Change in global left ventricular ejection fraction between initial examination at study entry and the 6 months follow up examination employing cardiac MRI | 6 months

SECONDARY OUTCOMES:
The application of 35 I.E./kg body weight erythropoetin beta s.c. once per week for 6 months is well tolerated and safe in patients after PCI. | 6 months
35 I.E. kg/KG erythropoetin beta s.c. once per week for 6 months improves left ventricular regional wall motion as assessed by cardiac MRI. | 6 months
35 I.E. kg/KG erythropoetin beta s.c. once per week for 6 months reduces serum levels of brain natriuretic peptide as a measure of heart failure. | 6 months
35 I.E. kg/KG erythropoetin beta s.c. once per week for 6 months improves peak VO2 as measured by spiroergometry | 6 months
35 I.E. kg/KG erythropoetin beta s.c. once per week for 6 months improves measures or cardiac diastolic dysfunction as assessed by echocardiography | 6 months
35 I.E. kg/KG erythropoetin beta s.c. once per week for 6 months improves cardiac tissue texture aqs assessed by contrast-enhanced cardiac MRI | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Martin W Bergmann, MD, Principal Investigator — Charité Camous Buch, University Medicine Berlin, Germany
Locations (2):
- Germany (2):
  - Charité Campus Buch, Berlin
  - Charité Campus Virchow, Berlin

REFERENCES:
- [Derived] Bergmann MW, Haufe S, von Knobelsdorff-Brenkenhoff F, Mehling H, Wassmuth R, Munch I, Busjahn A, Schulz-Menger J, Jordan J, Luft FC, Dietz R. A pilot study of chronic, low-dose epoetin-beta following percutaneous coronary intervention suggests safety, feasibility, and efficacy in patients with symptomatic ischaemic heart failure. Eur J Heart Fail. 2011 May;13(5):560-8. doi: 10.1093/eurjhf/hfr002. PMID 21505058